CLINICAL TRIAL: NCT00210028
Title: Open, Single-Arm Phase II Study Assessing Efficacy of ZARNESTRA™ Combined With Tamoxifen in Patients With Advanced or Metastatic Breast Cancer Expressing the Estrogen and/or Progesterone Receptor
Brief Title: Study Assessing Efficacy of ZARNESTRA™ Combined With Tamoxifen in Patients With Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03 SEIN 04
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Zarnestra; Tamoxifen; estrogen receptor; progesterone receptor
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; tipifarnib

INTERVENTIONS:
Drug: Tamoxifen
Drug: Zarnestra

SUMMARY:
The purpose of this study is to evaluate the objective response rate when ZARNESTRA is added to treatment with tamoxifen

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, metastatic or locally advanced inoperable breast cancer
* Tumor considered potentially hormone-sensitive, i.e. presence by IHC of hormone receptors for estrogens (ER+ for more than 10% of cells) and/or progesterone (Pg+ for more than 10% of cells) or both. This expression may have been detected on the primary tumor or at a metastatic site. The method used will be reassessed by IHC if it involves a radioligand technique whenever it is possible to obtain histological material.
* Progressing on treatment with tamoxifen, given either as adjuvant treatment or for advanced/metastatic breast cancer. Any previous treatment with a steroidal or nonsteroidal antiaromatase in a neo-adjuvant, adjuvant or metastatic situation is permitted. Likewise, any previous treatment with chemotherapy and/or herceptin in a nonmetastatic situation is permitted.
* Post-menopausal patients
* Age > 18 years
* At least one measurable lesion according to the Response Evaluation Criteria for Solid Tumors (RECIST) criteria; for patients who only have bone metastases, an evaluable non-irradiated lytic lesion is required
* Performance Status (WHO): PS ≤ 2 (Appendix 1).
* Laboratory tests in accordance with the following criteria:

Neutrophils ≥ 2x109/l,Platelets ≥ 100x109/l,Hemoglobin ≥ 10 g/dl, ASAT, ALAT ≤ 2.5 N , or < 5 N when liver metastasis,bilirubin ≤ 1.5 N creatinin ≤ 1.5 N

* Signed, written consent before any study-related procedure

Exclusion Criteria:

* Men
* Pre-menopausal patients who are not receiving concurrent LHRH agonist therapy
* ER- and PR-negative patients
* Contraindication to antiestrogens (thromboembolic risk) or ZARNESTRA
* Non metastatic tumor susceptible to management by radiotherapeutic and/or surgical means
* T4d inflammatory tumor (PEV 2 or 3).
* Short-term, life-threatening lesions: hepatic invasion > 1/3 of liver volume, pulmonary lymphangitis, uncontrolled cerebral metastases, carcinomatous meningitis
* Sensory neuropathy > or = grade 1 (WHO)
* Previous history of uncontrolled cancers or controlled for less than 5 years, except basal cell skin cancers and in situ cancers of the cervix.
* Chronic diseases (somatic or psychiatric) with a poor prognosis
* subjects with enzyme-inducing anti-convulsants (e.g., phenytoin, phenobarbital, carbamazepine) : this treatment is not permitted while taking ZARNESTRA
* Patients who, for family, social, geographic or psychological reasons, could not be followed up correctly.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-08; Study Completion 2008-08

PRIMARY OUTCOMES:
To evaluate the objective response rate when ZARNESTRA is added to administration of tamoxifen in patients suffering from metastatic or advanced inoperable breast cancer, who are progressing on tamoxifen treatment

SECONDARY OUTCOMES:
To evaluate the time to progression
To evaluate the clinical benefit (response + stable disease at 6 months)
To evaluate the safety of the combination ZARNESTRA and tamoxifen
To evaluate a possible pharmacokinetic interaction between ZARNESTRA and tamoxifen
To evaluate the biological predictive and prognostic factors of a response

CONTACTS AND LOCATIONS:
Overall Officials: Henri Roché, Pr, Principal Investigator — Institut Claudius Regaud
Locations (3):
- France (3):
  - Institut Bergonie, Bordeaux
  - Institut Val d'Aurelle_ Paul Lamarque, Montpellier
  - Institut Claudius Regaud, Toulouse